CLINICAL TRIAL: NCT06494540
Title: Prospective Non-interventional Study (NIS) to Examine the Effectiveness of Tremelimumab + Durvalumab + Platinum Chemotherapy (TDC) in Patients With Metastatic Non-squamous NSCLC and High-risk Genetic Alterations
Brief Title: NIS to Examine the Effectiveness of TDC in Patients With Metastatic Non-squamous NSCLC and High-risk Genetic Alterations
Acronym: NAUTIC
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D419MR00003
Record Dates: First submitted 2024-06-20; First posted 2024-07-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Non-squamous Metastatic Non-Small-Cell Lung Carcinoma
Keywords: NSCLC,; mNSCLC,; KRAS,; STK11,; KEAP1,; TP53,; POSEIDON,; Tremelimumab,; Durvalumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective, multicenter, non-interventional study (NIS) in Germany aims to collect real-life data of patients with non-squamous (NSQ) metastatic non-small cell lung cancer (mNSCLC) (incl. large cell neuroendocrine carcinoma (LCNEC) if considered NSCLC-like by the treating physician) for whom 1st line treatment initiation with tremelimumab and durvalumab in combination with a platinum-based chemotherapy (TDC) according to marketing authorization was scheduled. The study aims to describe the effectiveness with respect to mutations in Kirsten rat sarcoma viral oncogene homolog (KRAS), Serine/threonine kinase 11 (STK11), Kelch-like ECH-associated protein 1 (KEAP1), and Tumor protein p53 (TP53) as well as expression of Thyroid transcription factor 1 (TTF-1) and Programmed death-ligand 1 (PD-L1) in routine clinical practice. The generated data aims to deepen the understanding of optimal, biomarker-guided treatment strategies for NSQ mNSCLC in distinct subgroups with a high medical need.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Decision to start first-line (1L) treatment with TDC according to the current SmPCs
* Histologically or cytologically confirmed diagnosis of NSQ mNSCLC (incl. LCNEC if considered NSCLC-like by the treating physician)
* No sensitizing epidermal growth factor receptor (EGFR) mutations or anaplastic lymphoma kinase (ALK) alterations
* Molecular Next Generation Sequencing (NGS) panel as per institutional standard has been initiated (including the following genes: KRAS, STK11, KEAP1, and TP53)
* TTF-1 expression analysis has been initiated
* PD-L1 expression analysis has been initiated
* Women of childbearing potential must use effective contraception during treatment with durvalumab and for at least 3 months after the last dose of durvalumab
* Ability to understand the study concept
* Provision of signed informed consent form in accordance with applicable local provisions

Exclusion Criteria:

* Current participation in interventional clinical trials
* Contraindications according to current SmPCs
* Any active tumor other than metastatic NSCLC

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with a histologically or cytologically confirmed NSQ mNSCLC (incl. LCNEC if considered NSCLC-like by the treating physician), planned treatment initiation with TDC according to applicable Summary of product characteristics (SmPCs) within routine clinical practice and initiated molecular gene panel analysis (including KRAS, STK11, KEAP1, and TP53) as well as PD-L1 and TTF-1 expression analyses are eligible for enrolment.
  Eligible patients will be included into the study after and independently of the treating physician's treatment and diagnostic decisions but no later than 21 days after application of the first TDC treatment cycle.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Two-year real-world overall survival (rwOS) rate of patients with NSQ mNSCLC in the total study population | Time from patient's index date until death by any cause, up to 24 months
  rwOS rate (percentage of patients being alive derived by Kaplan-Meier methods) at 24 months in the total study population. Patients without a date of death will be censored at last activity in the database, or the end of the study period, whichever occurs first.
Two-year real-world overall survival (rwOS) rate of patients with NSQ mNSCLC in patients with mutations in KRAS | Time from patient's index date until death by any cause, up to 24 months
  rwOS rate (percentage of patients being alive derived by Kaplan-Meier methods) at 24 months in patients with mutations in KRAS. Patients without a date of death will be censored at last activity in the database, or the end of the study period, whichever occurs first.
Two-year real-world overall survival (rwOS) rate of patients with NSQ mNSCLC in patients with mutations in STK11 | Time from patient's index date until death by any cause, up to 24 months
  rwOS rate (percentage of patients being alive derived by Kaplan-Meier methods) at 24 months in patients with mutations in STK11. Patients without a date of death will be censored at last activity in the database, or the end of the study period, whichever occurs first.

SECONDARY OUTCOMES:
Real-world overall survival (rwOS) in the total study population | 6, 12 and 18 months
  rwOS rate (percentage of patients being alive derived by Kaplan-Meier methods) at 6, 12 and 18 months
Median overall survival (mOS) in the total study population | up to 24 months
  OS is defined as the time from the date of first documented dose of TDC until death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive. Median OS will be calculated using the Kaplan-Meier technique.
Real-world overall survival (rwOS) in a subgroup of patients with mutation in KRAS | 6, 12 and 18 months
  rwOS rate (percentage of patients being alive derived by Kaplan-Meier methods) at 6, 12 and 18 months
Median overall survival (mOS) in a subgroup of patients with mutation in KRAS | up to 24 months
  OS is defined as the time from the date of first documented dose of TDC until death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive. Median OS will be calculated using the Kaplan-Meier technique.
Real-world overall survival (rwOS) in a subgroup of patients with mutation in STK11 | 6, 12 and 18 months
  rwOS rate (percentage of patients being alive derived by Kaplan-Meier methods) at 6, 12 and 18 months
Median overall survival (mOS) in a subgroup of patients with mutation in STK11 | up to 24 months
  OS is defined as the time from the date of first documented dose of TDC until death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive. Median OS will be calculated using the Kaplan-Meier technique.
Real-world treatment response of TDC, as judged by the treating physician | up to 24 months
  Treatment response in terms of overall response rate (ORR), being defined as the proportion of patients with complete response (CR) or partial response (PR) as best overall response, CR or PR, at ≥1 visit during treatment with TDC.
Duration of response (DoR) | up to 24 months
  Duration of response (DoR), being defined as time from documented CR or PR until documentation of progressive disease (PD), or death by any cause will be analyzed with Kaplan-Meier methods. Patients without documentation of PD will be censored with their last date in the database known to be without PD, or the end of study date, whichever occurs first. Patients who received a subsequent line mNSCLC therapy after TDC before disease progression or death will be censored with the start date of this new therapy.
Real-world progression-free survival (rwPFS) | up to 24 months
  rwPFS is defined as time from patient's index date until first date of PD or death by any cause and will be analyzed by Kaplan-Meier methods.
Safety: Collection of Adverse Events (AE) | up to 24 months
  Safety evaluated based on type of Adverse Event (AE), intensity, causal relationship to treatment, duration, handling, outcome, and seriousness.

CONTACTS AND LOCATIONS:
Locations (21):
- Germany (21):
  - Research Site, Bad Homburg
  - Research Site, Berlin
  - Research Site, Celle
  - Research Site, Chemnitz
  - Research Site, Frankfurt
  - Research Site, Georgsmarienhütte
  - Research Site, Gera
  - Research Site, Goslar
  - Research Site, Halle-Dolau
  - Research Site, Hanover
  - Research Site, Herne
  - Research Site, Koln-Mehrheim
  - Research Site, Mainz
  - Research Site, Marburg
  - Research Site, Münnerstadt
  - Research Site, Neuss
  - Research Site, Ravensburg
  - Research Site, Treuenbrietzen
  - Research Site, Ulm
  - Research Site, Wiesbaden
  - Research Site, Zwickau

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca (AZ) group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/